CLINICAL TRIAL: NCT05607641
Title: A Multicenter, Randomized, Open-Label, Phase II/III Clinical Trial Evaluating the Efficacy and Safety of a Fixed Combination of Ketorolac / Pitofenone / Fenpiverinium Compared to Active Control in Patients With Pain After Surgical Abdominal and Pelvic Operations
Brief Title: Efficacy and Safety Study of Ketorolac / Pitofenone / Fenpiverinium for the Treatment of Patients With Pain After Surgical Abdominal and Pelvic Operations
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Darnitsa Pharmaceutical Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KPF07-T
Record Dates: First submitted 2022-10-27; First posted 2022-11-07 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Postsurgical Pain
Keywords: postsurgical pain; abdominal operation; pelvic operation; ketorolac tromethamine; pitofenone hydrochloride; fenpiverinium bromide
MeSH Terms: conditions — Pain, Postoperative | interventions — Ketorolac Tromethamine; Solutions

STUDY DESIGN:
Intervention Model Description: A prospective, multicenter, randomized, open-label, parallel-group comparative clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ketorolac tromethamine, solution for injection then Neospastil, film-coated tablets (Other)
  Interventions: Drug: Ketorolac tromethamine, solution for injection then Neospastil, film-coated tablets
- Ketorolac tromethamine, solution for injection then Ketorolac tromethamine, coated tablets (Active Comparator)
  Interventions: Drug: Ketorolac tromethamine, solution for injection then Ketorolac tromethamine, coated tablets
- Neospastil, solution for injection then Neospastil, film-coated tablets (Experimental)
  Interventions: Drug: Neospastil, solution for injection then Neospastil, film-coated tablets

INTERVENTIONS:
Drug: Ketorolac tromethamine, solution for injection then Neospastil, film-coated tablets — These medicines were used for patients of Group 1 (phase II) and Group 4 (phase III).
  Stage 1 (1st day of study treatment) - Ketorolac tromethamine, solution for injection, 1 ml every 8 hours.
  Stage 2 (2nd day of study treatment) - Neospastil, film-coated tablets, 1 tablet every 6 hours.
  Stage 3 (3rd-5th days of study treatment) - Neospastil, film-coated tablets, 1 tablet on demand with an interval of at least 6 hours, not more than 4 tablets per day.
  Arms: Ketorolac tromethamine, solution for injection then Neospastil, film-coated tablets
Drug: Ketorolac tromethamine, solution for injection then Ketorolac tromethamine, coated tablets — These medicines were used for patients of Group 2 (phase II) and Group 5 (phase III).
  Stage 1 (1st day of study treatment) - Ketorolac tromethamine, solution for injection, 1 ml every 8 hours.
  Stage 2 (2nd day of study treatment) - Ketorolac tromethamine, coated tablets, 1 tablet every 6 hours.
  Stage 3 (3rd-5th days of study treatment) - Ketorolac tromethamine, coated tablets, 1 tablet on demand with an interval of at least 6 hours, not more than 4 tablets per day.
  Arms: Ketorolac tromethamine, solution for injection then Ketorolac tromethamine, coated tablets
Drug: Neospastil, solution for injection then Neospastil, film-coated tablets — These medicines were used for patients of Group 3 (phase II) and Group 6 (phase III).
  Stage 1 (1st day of study treatment) - Neospastil, solution for injection, 2 ml every 8 hours.
  Stage 2 (2nd day of study treatment) - Neospastil, film-coated tablets, 1 tablet every 6 hours.
  Stage 3 (3rd-5th days of study treatment) - Neospastil, film-coated tablets, on demand 1 tablet with an interval of at least 6 hours, not more than 4 tablets per day.
  Arms: Neospastil, solution for injection then Neospastil, film-coated tablets

SUMMARY:
Neospastil (ketorolac tromethamine / pitofenone hydrochloride / fenpiverinium bromide fixed-dose combination) in a form of solution for injections and film-coated tablets has been studied as a treatment for pain after surgical abdominal and pelvic operations. The aim of the study was to test the hypothesis that Neospastil was non-inferior (phase II) and superior (phase III) than ketorolac tromethamine monotherapy due to the additional relaxing effect of pitofenone and fenpiverinium on the smooth muscles of internal organs. The study also aimed to show that Neospastil is safe and well-tolerated in people who have pain after surgical abdominal and pelvic operations. Study treatment was initiated with parenteral form of study drug (first 24 hours) and then switched to oral formulation. This trial was conducted in accordance with the ethical principles of Good Clinical Practice and International Council for Harmonization (ICH) Harmonized Tripartite Guidelines.

ELIGIBILITY:
Criteria Abbreviations: New York Heart Association (NYHA).

Inclusion Criteria:

1. Age of 18-64 years inclusive and body weight of ≥ 50 kg.
2. The estimated need to use the first dose of the IMP no later than 8 hours after the completion of minimally invasive surgical abdominal and pelvic operations.
3. Immediately before randomization, there is a moderate to severe pain associated with minimally invasive surgical abdominal and pelvic operation (the overall assessment of pain at rest is 4-8 points inclusively in 11-point NRS).
4. At the time of minimally invasive surgery, the patient's condition corresponded to the class I-III of general anesthesia risk according to the classification of the American Society of Anesthesiologists (ASA).
5. The patient is able to adequately assess his/her condition and fill in yourself the patient's diary.
6. The patient agrees to participate in the clinical trial and fulfill all the requirements of the trial and has signed the informed consent form.
7. According to the investigator, IMP is an adequate tactic for postoperative analgesia.

Exclusion Criteria:

1. Hypersensitivity or allergic reactions/conditions associated with ketorolac, pitofenone, fenpiverinium, any other components of IMPs, acetylsalicylic acid or other non-steroidal anti-inflammatory drugs.
2. The patient has another disease/condition that requires constant use of non-topical analgesics and/or anti-inflammatory agents or, in the opinion of the investigator, disturbs the patient's perception of postoperative pain.
3. The need for postoperative treatment in the intensive care unit for any reason.
4. Active peptic ulcer, recent gastrointestinal bleeding or perforation, history of peptic ulcer or gastrointestinal bleeding.
5. History of bronchial asthma.
6. Severe heart failure (class III-IV according to NYHA).
7. Severe liver failure (including an increase in the activity of alanine aminotransferase and/or aspartate aminotransferase in the blood more than three times the upper limit of normal).
8. Moderate to severe renal failure (blood creatinine concentration > 160 μmol/l).
9. Suspected or confirmed cerebrovascular bleeding, hemorrhagic diathesis, including blood coagulation disorders and high risk of bleeding.
10. Dehydration with the risk of kidney failure due to a decrease in the volume of circulating blood.
11. Benign prostatic hyperplasia of the ΙΙ and ΙΙΙ degree.
12. Cardiovascular diseases in which an increase in heart rate may be undesirable (for example, atrial fibrillation, tachycardia [pulse rate at rest > 100 bpm], severe arterial hypertension), as well as an artificial pacemaker.
13. Glaucoma.
14. Signs of intestinal obstruction and/or history of megacolon.
15. Anemia (hemoglobin concentration < 90 g/l) and/or leukopenia (leukocyte count < 3.2x109/l) according to the results of preoperative laboratory examination.
16. Diseases or conditions that make it impossible to take drugs orally in accordance with the Clinical Trial Protocol and/or disrupt their absorption in the gastrointestinal tract.
17. The use of drugs prohibited by the Clinical Trial Protocol before the start of study treatment and/or the need to use drugs prohibited by the Clinical Trial Protocol during the investigational treatment.
18. Mental disorder/illness, which, in the opinion of the investigator, may prevent the patient from fulfilling all the requirements of the trial.
19. Pregnancy or lactation.
20. Within 30 days prior to randomization, the use of a drug or medical product in another clinical trial.
21. The patient has already been previously randomized in this trial.

Criteria to start the 2nd stage of treatment, the patient had to meet the criteria for switching to IMP for oral administration:

* pain level of 4-6 points at movements according to the 11-point Numerical Rating Scale (NRS) (7 points were allowed, if pain level at rest did not exceed 6 points according to 11-point NRS);
* no more than 12 hours have passed since the last use of IMP;
* oral analgesic use is an adequate tactic for postoperative analgesia.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 424 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2022-05-07 (Actual); Study Completion 2022-05-13 (Actual)

PRIMARY OUTCOMES:
Proportion of study subjects who achieved a response to treatment within the first 24 hours of using IMP in the form of solution for injections. | Stage 1 (1st day of treatment).
  This primary endpoint was evaluated using the following combined primary (main) efficacy variable.
  The patient who met all of the following criteria (1.1-1.3) was considered as a "responder". The patient who didn't meet at least one of the following criteria was classified as a "non-responder".
  1.1. Reduction in pain intensity at rest compared to the initial level by ≥ 50 % within the first 90 min. after the first dose of IMP in the form of a solution for injections (i.e., at least at one of the following time points 30 [±5] min., 60 [±10] min. and/or 90 [±15] min.).
  1.2. During the study treatment, the intensity of pain at rest is < 4 points on the 11-point NRS at time points between 2 and 24 hours (i.e. 120 [±20] min., 4 [±0.5] h., 6 [±1] h., 8 [±1] h., 16 [±2] h. and 24 [±2] h.) after starting the use of IMP in the form of solution for injections.
  1.3. The study subject didn't receive other analgesics during the first 24 hours of the study treatment.
Proportion of study subjects who achieved a response to treatment within the first 24 hours of using IMP in the form of tablets. | Stage 2 (2nd day of treatment).
  This primary endpoint was evaluated using the following combined primary (main) efficacy variable.
  The patient who met all of the following criteria (2.1-2.3) was considered as a "responder". The patient who didn't meet at least one of the following criteria was classified as a "non-responder".
  2.1. Reduction in pain intensity at movements compared to the initial level by ≥ 50 % within the first 120 min. after the first dose of IMP in the form of tablets (i.e., at least at one of the following time points 60 [±10 min., 90 [±15] min. and/or 120 [±20] min.).
  2.2. During the study treatment, the intensity of pain during movement is < 4 points on the 11-point NRS at time points between 3 and 24 hours (i.e. 3 [±0.5] h, 4 [±0.5] h, 6 [±1] h, 12 [±2] h, 18 [±2] h and 24 [±2] h) after starting to use IMP in the form of tablets.
  2.3. The study subject didn't receive other analgesics within 24 hours since beginning of the IMP usage in the form of tablets.

SECONDARY OUTCOMES:
Time to a noticeable and distinct decrease in the intensity of pain at rest from the first dose of IMP in the form of a solution for injections. | Stage 1 (1st day of treatment)
Pain intensity at rest and during movements according to the 11-point NRS at time points during the study treatment. | Stage 1 (1st day of treatment), Stage 2 (2nd day of treatment) and Stage 3 (3rd-5th days of treatment)
Area under the curve of pain intensity at rest and during movements according to the 11-point NRS at time points within 24 hours after the first dose of IMP in the form of solution for injections and IMP in the form of tablets. | Stage 1 (1st day of treatment) and Stage 2 (2nd day of treatment)
Sum of pain intensity differences (SPID) at rest and during movements within 6 hours after the first dose of IMP in the form of solution for injections or IMP in the form of tablets. | First 6 hours of Stage 1 (1st day of treatment) and Stage 2 (2nd day of treatment)
The proportion of patients who achieved a response to treatment. | Stage 1 (1st day of treatment), Stage 2 (2nd day of treatment) and Stage 3 (3rd-5th days of treatment)
  A response to treatment based on the patient's overall assessment of pain control within 24 hours using of IMP in the form of a solution for injections and IMP in the form of tablets, as well as at the end of the study treatment.
The number of IMP doses administered during 3-5 days of the study treatment (per patient). | Stage 3 (3rd-5th day of treatment)
Proportion of patients who used another analgesic since the first dose of IMP. | Stage 1 (1st day of treatment), Stage 2 (2nd day of treatment) and Stage 3 (3rd-5th days of treatment)

CONTACTS AND LOCATIONS:
Locations (14):
- Ukraine (14):
  - Regional municipal nonprofitable institution "Chernivtsi regional clinical hospital", urological department, Chernivtsi
  - Communal enterprise "Dnipropetrovsk Regional Clinical Hospital named after І.І. Mechnikov" Dnipropetrovsk Regional Council", urology department №1, Dnipro
  - Communal enterprise "Dnipropetrovsk Regional Clinical Hospital named after І.І. Mechnikov" Dnipropetrovsk Regional Council", urology department №2, Dnipro
  - Communal noncomercial enterprise of the Kharkiv Regional Council "Regional Medical Clinical Center of Urology and Nephrology named after V.I. Shapovala", urology department №5, Kharkiv
  - Communal noncomercial enterprise "Kyiv City Clinical Hospital #3" Kyiv City Council (Kyiv City State Administration), urological department, Kyiv
  - Medical Center of the LLC "Harmony of Beauty", Kyiv
  - State Institution "Institute of Urology of the National Academy of Medical Sciences of Ukraine", I Urological Department, Kyiv
  - Communal noncomercial enterprise of the Lviv Regional Council "Lviv Regional Clinical Hospital", department of urology, Lviv
  - Municipal Non-profit Enterprise "Lviv Clinical Hospital for Emergency Medical Care", Lviv
  - Communal noncomercial enterprise "City Clinical Hospital #10" Odesa City Council, urological department #2, Odesa
  - Medical-diagnostic center" Zakarpattya center of surgical innovations" Astra-med "of limited liability company" Clinic of healthy family "Astramed", Uzhhorod
  - Communal noncomercial enterprise" Vinnytsia City Clinical Hospital" Mother and Child Center", department of gynecology with minimally invasive operations, Vinnytsia
  - Limited Liability Company "Innomed Center of Endosurgery", Vinnytsia
  - Communal noncomercial enterprise "City Hospital of Emergency and Ambulance" of Zaporizhia City Council, Department of Surgery with the Center for Gastrointestinal Bleeding, Zaporizhzhya

IPD SHARING:
Plan to Share IPD: No